CLINICAL TRIAL: NCT01318655
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of NKTR-118 Following Single and Multiple Ascending Oral Dose Administration in Healthy Young and Elderly Japanese Subjects, and an Open Randomized, Crossover Study to Investigate the Effect of Food on the Pharmacokinetics After Single Oral Doses of NKTR-118 in Healthy Male Japanese Subjects
Brief Title: Single and Multiple Ascending Dose Study for NKTR-118 and Cross-over Study to Investigate the Effect of Food for NKTR-118 in Japanese Healthy Subjects
Acronym: Japan SMAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D3820C00020
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Last update posted 2011-08-25 (Estimated); Status verified 2011-08

CONDITIONS: Healthy
Keywords: Phase I; Japan; SAD; MAD
MeSH Terms: interventions — naloxegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NKTR-118 (Experimental)
  Interventions: Drug: NKTR-118
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NKTR-118 — Tablet, Oral, Once daily
  Arms: NKTR-118
Drug: Placebo — Tablet, Oral, Once daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of NKTR-118 with healthy subjects.

DETAILED DESCRIPTION:
A Phase I, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of NKTR-118 following single and multiple ascending oral dose administration in healthy young and elderly Japanese subjects, and an Open Randomized, Crossover Study to Investigate the Effect of Food on the Pharmacokinetics after single oral doses of NKTR-118 in healthy male Japanese subjects

ELIGIBILITY:
Inclusion Criteria:

* 20 Years to 45 Years, 65 Years to 80 Years
* Body mass index (BMI): 18 to 27 kg/m
* Male subjects should be willing to use barrier contraception ie, condoms, from the day of dosing until 3 months after dosing with the investigational product.
* Non-smokers or ex-smokers (not smoked in the past 3 months).

Exclusion Criteria:

* Clinically relevant disease and/or abnormalities (past or present)
* Clinically relevant abnormalities in physical examinations,vital signs,clinical chemistry, hematology or urinalysis as judged by the investigator
* Use of any prescribed or non-prescribed medication including herbal remedies, vitamins and minerals during the two weeks prior to the first administration of investigational product

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Investigate the safety and tolerability of NKTR-118 using incidence of Adverse Events

SECONDARY OUTCOMES:
Assessment of drug concentrations in plasma by characterizing PK parameters (AUC)
Assessment of drug concentrations in plasma by characterizing PK parameters (Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sostek, MD, Study Director — AstraZeneca; Shunji Matsuki, MD, Principal Investigator — Kyusyu Clinical Phramacology Research Clinic; Yukiya Sasaki, MD, Principal Investigator — AstraZeneca
Locations (1):
- Research Site, Chūōku, Fukuoka, Japan